CLINICAL TRIAL: NCT05541523
Title: Does Cognitive Behavioural Therapy or Mindfulness-based Therapy Improve Mental Health and Emotional Labor Among Nurses Who Care the End-of-life Patients? A Randomized Controlled Trial
Brief Title: Improve Mental Health and Emotional Labor Among Nurses Who Care the End-of-life Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Huichao Zhang (Other)
Responsible Party: Sponsor-Investigator, Huichao Zhang, Professor, Nanjing University of Traditional Chinese Medicine
Organization: Nanjing University of Traditional Chinese Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SJCX22_0702
Record Dates: First submitted 2022-09-12; First posted 2022-09-15 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: End-of-life; Depression, Anxiety
MeSH Terms: conditions — Death; Depression; Anxiety Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cognitive behavioural therapy (Experimental)
  Interventions: Behavioral: mindfulness-based therapy
- mindfulness-based therapy (Experimental)
  Interventions: Behavioral: cognitive behavioural therapy

INTERVENTIONS:
Behavioral: cognitive behavioural therapy — The three therapists in the cognitive behavioural group therapy condition were two students of master's degree of nursing with formal education in cognitive therapy and one psychological specialist nurse working in a palliative care unit. There was no evidence of significant deviation from the protocol.
  Arms: mindfulness-based therapy
Behavioral: mindfulness-based therapy — The two therapists in the mindfulness-based stress reduction condition were one clinical psychologist and one student of master's degree of nursing with formal education in mindfulness.Both interventions were manualized. To assure adherence to the study protocol meetings between the therapists and the researchers were organized regularly and the therapists detailed the content of each group session in clinical records which were frequently monitored by a research assistant.
  Arms: cognitive behavioural therapy

SUMMARY:
CBT: cognitive behavioural therapy MBT: mindfulness-based therapy

DETAILED DESCRIPTION:
Nurses caring for terminally ill patients suffer from negative emotions and emotional labor, which may lead to a decline in the quality of end-of-life care. CBT and MBT are currently two commonly used psychological methods. They can be effective in improving bad mood. However, to the best of our knowledge, no investigators have used CBT and MBT among nurses caring for terminally ill patients. Could CBT and MBT be effective in alleviating the psychological distress of these nurses? Which psychological method is more effective?

ELIGIBILITY:
Inclusion Criteria:

* (1) Eligible participants were the nurses who nursing patients with stage IV cancer or other incurable diseases;
* (2) agree to participate in this research;
* (3) no history of mental illness.

Exclusion Criteria:

* None

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Anxiety | up to 8 weeks
  The Hamilton Anxiety Rating Scale (HAM-A), developed by Hamilton in 1959,26 was used in this study to assess the anxiety level of the patients. The HAM-A contains 14 items, each scored on a 5-point scale (0, asymptomatic; 1, mild symptoms; 2, moderate symptoms; 3, severe symptoms; 4, extremely severe symptoms). The total sum score, ranging from 0 to 56, can be classified into four levels: 0, no anxiety symptoms; 1-17, mild anxiety; 18-24, moderate anxiety; 25-56, severe anxiety.
Emotional labor | up to 8 weeks
  Chinese version scale of emotional labor(C-ELS). Permission to use the Chinese version of the instruments was obtained. To the best of our knowledge, this is the first time these questionnaires are used in palliative care programs in China, using a five-point Likert type scale ("1" = "strongly disagree," "7" = "strongly agree"). The scale divided emotional labor into four part surface acting, deep acting, expression of naturally felt emotions and emotion termination. The Cronbach's α of surface acting, deep acting, expression of naturally felt emotions and emotion termination were 0.714, 0.743, 0.846, 0.758, respectively.
Self-Efficacy | up to 8 weeks
  Occupational Coping Self-Efficacy Scale for Nurses ( OCSE-N, Occupational Coping Self-Efficacy Scale for Nurses ), a total of 9 items, using Likert 5-level scoring method, 1 means ' can not easily deal with ' to 5 means ' can easily deal with ', the total score range of 9 to 45 points, the higher the score, the higher the occupational coping self-efficacy of nurses.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - the First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Wu Ye, Nanjing, Jiangsu

IPD SHARING:
Plan to Share IPD: No